CLINICAL TRIAL: NCT02458157
Title: Forced Fluid Removal vs. Usual Intensive Care in High-risk Acute Kidney Injury With Severe Fluid Overload - A Randomized Controlled Trial
Brief Title: Forced Fluid Removal in High Risk Acute Kidney Injury
Acronym: FFAKI
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Very low recruitment rates
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Aalborg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FFAKI; 2015-001701-13 (EudraCT Number)
Record Dates: First submitted 2015-05-21; First posted 2015-06-01 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Acute Kidney Injury; Fluid Overload; Critical Illness
Keywords: ICU; Intensive; CRRT; Fluid Removal; AKI; Critical Care
MeSH Terms: conditions — Acute Kidney Injury; Edema; Critical Illness | interventions — Furosemide; Continuous Renal Replacement Therapy; Resuscitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Forced Fluid Removal (Experimental): The experimental intervention is guided by a therapeutic goal of average negative fluid balance ≥ 1 ml/kg/h and safety variables indicating inadequate circulation (lactate ≥ 4, MAP < 50 or mottling beyond the edge of kneecaps).
  The effect of fluid removal is evaluated three times daily (06:00. 14:00 and 22:00), while the safety variables are evaluated continuously. Resuscitation is started if one or more signs of inadequate circulation is present.
  The first choice for fluid removal is diuretic therapy with furosemide, which is continued for a minimum of 8 hours. If the therapeutic goal (negative fluid balance ≥ 1 ml/kg/h) is not achieved and/or maintained by furosemide alone, then fluid removal with continuous renal replacement therapy (CRRT) is initiated.
  Interventions: Drug: Furosemide (Furix); Other: Continuous renal replacement therapy (CRRT); Other: Resuscitation
- Usual Care (Active Comparator): Usual Care at the discretion of the treating clinicians, except for the initiation of renal replacement therapy (RRT).
  Interventions: Other: Usual Care

INTERVENTIONS:
Drug: Furosemide (Furix) — * Loading dose: 40 mg I.V.
  * Infusion rate 40 mg/h
  * Continued until neutral cumulative fluid balance is achieved (the overall treatment goal) or average negative fluid balance is below 1 ml/kg/h for 8 hours.
  Other Names: Furix
  Arms: Forced Fluid Removal
Other: Continuous renal replacement therapy (CRRT) — * Initiated in case of contraindications or inadequate effect of furosemide.
  * Fluid removal is started at 2 ml/kg/h
  * The efficacy is evaluated 3 times daily and removal rate increased by 0.5 ml/kg/h if the therapeutic goal is not achieved
  Other Names: CRRT
  Arms: Forced Fluid Removal
Other: Resuscitation — The physiologic response to fluid removal is monitored with three variables indicating inadequate circulation. These are:
  * Mottling beyond the edge of kneecaps
  * Hypotension (MAP < 50) resistant to inotropes and vasopressors
  * Plasma lactate ≥ 4 mmol/l
  Mottling and MAP are monitored continuously and lactate is measured routinely 4-6 times each day and on clinical indication. If one or more variable is present:
  1. Fluid removal is paused
  2. A crystalloid fluid bolus of 250-500 ml is given
  3. Circulatory status is reevaluated within 30 minutes
  4. Step 1-3 is repeated until signs of inadequate circulation have been resolved for minimum 1 hour
  5. Fluid removal is restarted in 25% reduced dose for minimum 4 hours before evaluation of effect.
  Arms: Forced Fluid Removal
Other: Usual Care — All interventions are performed at the discretion of the treating physician apart from initiation of renal replacement therapy which is discouraged unless one or more of the following criteria are met:
  * Hyperkalaemia (p-K+ > 6 mmol/l)
  * Severe metabolic acidosis attributable to AKI (pH < 7.25 and standard base excess < -10 mmol/l) resistant to IV bicarbonate infusion
  * Severe respiratory failure with PaO2/FiO2 < 13 kPa and bilateral infiltrates/oedema on the chest x-ray.
  * Progressive azotaemia and a blood urea nitrogen (BUN) > 25 mmol/l.
  Arms: Usual Care

SUMMARY:
The objective of this pilot trial is to assess the feasibility of forced fluid removal in patients admitted to the intensive care unit (ICU) with high-risk AKI and severe fluid overload. The intervention will use furosemide infusion and/or continuous renal replacement therapy (CRRT) to achieve and maintain a neutral cumulative fluid balance. The intervention will be compared to standard of care as reflected in the kidney disease improving global outcome (KDIGO) guidelines.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common and serious complication in patients admitted to ICU. A core element of critical care is resuscitation with crystalloid solutions. In many cases fluid accumulates and patients become fluid overloaded (positive fluid balance > 10% of bodyweight). This is especially true in patients with AKI, since they often have impaired ability to excrete salt and water. Most observational suggests harm with increased positive fluid balance.

Objectives: To assess feasibility of forced fluid removal with diuretics and/or CRRT in ICU patients with AKI and severe fluid overload, compared to current clinical practice.

Design: Multicentre, parallel group, randomized, assessor blinded pilot-trial with adequate generation of allocation sequence, and allocation concealment.

Trial Size: The pilot study is planned to include 50 patients. Inclusion is expected to start in August 2015.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Acute Kidney Injury defined according to the KDIGO criteria
* Renal Recovery Score ≤ 60%. (Calculated using www.renal-recovery-score.com)
* Fluid overload defined as a positive fluid balance ≥ 10% of ideal body weight.
* Able to undergo randomization within 12 hours of fulfilling other inclusion criteria

Exclusion Criteria:

* Known pre-hospitalization advanced chronic kidney disease. (eGFR < 30 mL/minute/1.73 m2 or chronic RRT.)
* Severe hypoxic respiratory failure (use of invasive ventilation and FiO2 > 80% and PEEP > 10 cm H2O)
* Severe burn injury (≥ 10% TBSA)
* Severe hypo- or hyper- natremia (< 120 or > 155 mmol/l)
* Hepatic coma
* Mentally disabled undergoing forced treatment
* Pregnancy/breast feeding
* Lack of commitment for on-going life support including RRT
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-10; Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

PRIMARY OUTCOMES:
Cumulative fluid balance | 5 days
  Calculated as the sum of daily intake - daily output, as registered on the daily ICU observation charts.

SECONDARY OUTCOMES:
Cumulative fluid balance | ICU stay expected average of 10 days
  participants will be followed for the duration of ICU stay, an expected average of 10 days
Mean daily fluid balance | ICU stay expected average of 10 days
  participants will be followed for the duration of ICU stay, an expected average of 10 days
Major protocol violations | ICU stay expected average of 10 days
  participants will be followed for the duration of ICU stay, an expected average of 10 days
Time to neutral cumulative fluid balance | 90 days
  No. of days until neutral cumulative fluid balance is achieved. Participants will be followed until neutral fluid balance is achieved or they reach the end of the observation period (90 days)
Accumulated serious adverse reactions | 90 days
  Serious adverse reactions related to fluid removal(atrial fibrillation, ischemic events and organ failure), furosemide (severe electrolyte disturbance, severe thrombocytopenia, hearing loss agranulocytosis and allergic reactions) and the infusion of noradrenaline (cerebral hemorrhage, cardiac arrhythmia, psychiatric symptoms) will be examined

OTHER OUTCOMES:
All cause mortality | 90 days
Days alive and out of hospital | 90 days
Days alive and out of mechanical ventilation | 90 days
Days alive and out of renal replacement therapy | 90 days
Renal recovery | 90 days
  Defined as 5 consecutive days of:
  * No renal replacement therapy
  * serum creatinine ≤ 150 % baseline value

CONTACTS AND LOCATIONS:
Overall Officials: Morten H Bestle, MD, Ph D, Principal Investigator — Nordsjællands Hospital. Dept. of Anaesthesiology and Intensive Care.; Anders Perner, Md, Ph D, Study Chair — Rigshospitalet. ITA 4131 / Dept of Intensive Care; Jens-Ulrik Jensen, MD, Ph D, Study Chair — Rigshospitalet, University of Copenhagen CHIP, Department of Infectious Diseases and Rheumatology, Section 2100; Michael Ibsen, MD, Ph D, Study Chair — Nordsjællands Hospital. Dept. of Anaesthesiology and Intensive Care.; Rasmus E Berthelsen, MD, Study Chair — Nordsjællands Hospital. Dept. of Anaesthesiology and Intensive Care.
Locations (3):
- Denmark (3):
  - Aalborg Universitetshospital, Anæstesi og intensiv afdeling, Aalborg
  - Nordsjællands Hospital. Dept. of Anaesthesiology and Intensive Care., Hillerød
  - Rigshospitale. ITA 4131 / Dept. of intensive care, København Ø

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Berthelsen RE, Perner A, Jensen AK, Rasmussen BS, Jensen JU, Wiis J, Behzadi MT, Bestle MH. Forced fluid removal in intensive care patients with acute kidney injury: The randomised FFAKI feasibility trial. Acta Anaesthesiol Scand. 2018 Aug;62(7):936-944. doi: 10.1111/aas.13124. Epub 2018 Apr 17. PMID 29664109
- [Derived] Berthelsen RE, Itenov T, Perner A, Jensen JU, Ibsen M, Jensen AEK, Bestle M. Forced fluid removal versus usual care in intensive care patients with high-risk acute kidney injury and severe fluid overload (FFAKI): study protocol for a randomised controlled pilot trial. Trials. 2017 Apr 24;18(1):189. doi: 10.1186/s13063-017-1935-2. PMID 28438182